CLINICAL TRIAL: NCT03916003
Title: Reducing the Risk of P. Vivax After Falciparum Infections in Co-endemic Areas - a Randomized Controlled Trial
Brief Title: Reducing the Risk of P. Vivax After Falciparum Infections in Co-endemic Areas
Acronym: PRIMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Tribhuvan University, Nepal (Other); Arba Minch University (Other); Addis Ababa University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-3288
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Malaria; Vivax Malaria; Falciparum Malaria
MeSH Terms: conditions — Malaria; Malaria, Vivax; Malaria, Falciparum | interventions — Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PQ7 (Experimental): high dose primaquine regimen over 7 days (1.0 mg/kg/day for 7 days)
  Interventions: Drug: primaquine
- standard care (No Intervention): As per national guidelines for P. falciparum treatment

INTERVENTIONS:
Drug: primaquine — Primaquine regimen over 7 days (1.0 mg/kg/day for 7 days)
  Arms: PQ7

SUMMARY:
This study is designed as a multi-centre randomized, open label trial to compare the safety and efficacy of a high dose primaquine (PQ) treatment in G6PD normal patients with P. falciparum to reduce the risk of subsequent P. vivax episodes to current standard practice of providing only schizontocidal treatment.

DETAILED DESCRIPTION:
Plasmodium vivax forms dormant liver stages that reactivate weeks or months following an acute infection. Recurrent infections can be associated with a febrile illness, a cumulative risk of severe anaemia, direct and indirect mortality, and are the most important source of onward transmission of the parasite. In co-endemic areas, there is a very high risk (up to 50%) of patients representing with P. vivax malaria following treatment of P. falciparum. Hence, in co-endemic regions there is a strong rationale for eradicating P. vivax hypnozoites from the liver in patients presenting with uncomplicated P. falciparum infections.

The recently completed multicentre IMPROV study compared the efficacy of a 7 day primaquine regimen (1.0 mg/kg/day for 7 days) with a 14 day regimen (0.5 mg/kg/day for 14 days). The 7 day PQ regimen was non-inferior to the 14 day regimen and 5-fold more efficacious at reducing P. vivax recurrence than the control.

This study is designed as a multicentre randomized, open label trial to compare the safety and efficacy of a high dose PQ treatment in G6PD normal patients with P. falciparum to reduce the risk of subsequent P. vivax episodes to current standard practice of providing only schizontocidal treatment.

ELIGIBILITY:
Inclusion Criteria:

* P. falciparum mono-infection
* Fever (axillary temperature ≥37.5⁰C) or history of fever in preceding 48 hours
* Age >1 years (≥ 18 years at the Ethiopia site)
* G6PD normal as defined by the Biosensor (SD Biosensor, ROK) at ≥70% of the adjusted male median (AMM) for each site
* Written informed consent
* Able to comply with all study procedures and timelines

Exclusion Criteria:

* General danger signs or symptoms of severe malaria
* Anaemia, defined as Hb <8g/dl
* Pregnant women as determined by Urine β-HCG pregnancy test
* Breast feeding women
* Known hypersensitivity to any of the drugs given
* Regular use of drugs with haemolytic potential
* Blood transfusion within the last 4 months

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2019-08-18 (Actual); Primary Completion 2022-05-14 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Incidence risk of any P. vivax parasitaemia at day 63 | 63 days
  The incidence risk of any P. vivax parasitaemia at day 63

SECONDARY OUTCOMES:
Incidence risk of symptomatic P. vivax parasitaemia at day 63 | 63 days
  incidence risk of symptomatic P. vivax parasitaemia at day 63
Incidence risk of all any P. vivax parasitaemia at day 28 and 42 | 28 and 42 days
  Incidence risk of all any P. vivax parasitaemia at day 28 and 42
Incidence risk of any P. falciparum malaria at day 28, 42 and 63 | 28/42/63 days
  incidence risk of any P. falciparum malaria at day 28, 42 and 63
proportion of patients vomiting their medication within 1 hour of administration | 1 hour
  proportion of patients vomiting their medication on the day of enrollment within 1 hour of administration
proportion of patients vomiting any of their PQ doses within 1 hour of administration | 7 days
  proportion of patients vomiting any of their PQ doses within 1 hour of administration
proportion of adverse events and serious adverse events | 63 days
  proportion of adverse events and serious adverse events
incidence risk of severe anaemia (Hb<5g/dl) and moderately severe anaemia (<7g/dl) and/or the risk for blood transfusion between day 3 and 7 | 7 days
  incidence risk of severe anaemia (Hb<5g/dl) and moderately severe anaemia (<7g/dl) and/or the risk for blood transfusion between day 3 and 7
• The incidence risk of ≥25% fall in haemoglobin since baseline with and without hemoglobinuria at day 3 and day 7 | 7 days
  • The incidence risk of ≥25% fall in haemoglobin since baseline with and without hemoglobinuria at day 3 and day 7
The incidence risk of ≥25% fall in haemoglobin to under 7g/dl with and without hemoglobinuria at day 3 and day 7 | day 7
  The incidence risk of ≥25% fall in haemoglobin to under 7g/dl with and without hemoglobinuria at day 3 and day 7
Incidence risk of P. falciparum gametocytaemia between day 7 and 63 | 63 days
  Incidence risk of P. falciparum gametocytaemia between day 7 and 63
Parasite clearance on day 1, 2 and 3 | 3 days
  Parasite clearance on day 1, 2 and 3
Fever clearance on day 1, 2 and 3 | 3 days
  Fever clearance on day 1, 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Kamala Thriemer, MD, Principal Investigator — Menzies School of Health Research
Locations (3):
- Icddrb, Upazila, Bangladesh
- Arba Minch University, Arba Minch, Ethiopia
- Puskesmas Mangili, Dusun Tenggara, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Statistical Analysis Plan will be made available to others. Data collected for the study, including individual patient data and the final trial dataset are reserved for the chief investigator and co-investigators of the trial. The trial will be reported in accordance with the Consolidated Standards of Reporting Trials (CONSORT) guidelines. Trial results will be published in peer-reviewed open access journals and disseminated to trial stakeholders, including participants, as per ethical guidelines.
Supporting Information: Study Protocol, SAP
Access Criteria: The data are available for access via the WorldWide Antimalarial Resistance Network (WWARN.org). Requests for access will be reviewed by a Data Access Committee to ensure that use of data protects the interests of the participants and researchers according to the terms of ethics approval and principles of equitable data sharing. Requests can be submitted by email to malariaDAC@iddo.org via the Data Access Form available at WWARN.org/accessing-data. The WWARN is registered with the Registry of Research Data Repositories (re3data.org).
URL: http://WWARN.org/accessing-data

REFERENCES:
- [Derived] Thriemer K, Degaga TS, Christian M, Alam MS, Rajasekhar M, Ley B, Hossain MS, Kibria MG, Tego TT, Abate DT, Weston S, Mnjala H, Rumaseb A, Satyagraha AW, Sadhewa A, Panggalo LV, Ekawati LL, Lee G, Anose RT, Kiros FG, Simpson JA, Karahalios A, Woyessa A, Baird JK, Sutanto I, Hailu A, Price RN. Primaquine radical cure in patients with Plasmodium falciparum malaria in areas co-endemic for P falciparum and Plasmodium vivax (PRIMA): a multicentre, open-label, superiority randomised controlled trial. Lancet. 2023 Dec 2;402(10417):2101-2110. doi: 10.1016/S0140-6736(23)01553-2. Epub 2023 Nov 15. PMID 37979594
- [Derived] Thriemer K, Degaga TS, Christian M, Alam MS, Ley B, Hossain MS, Kibria MG, Tego TT, Abate DT, Weston S, Karahalios A, Rajasekhar M, Simpson JA, Rumaseb A, Mnjala H, Lee G, Anose RT, Kidane FG, Woyessa A, Baird K, Sutanto I, Hailu A, Price RN. Reducing the risk of Plasmodium vivax after falciparum infections in co-endemic areas-a randomized controlled trial (PRIMA). Trials. 2022 May 18;23(1):416. doi: 10.1186/s13063-022-06364-z. PMID 35585641